CLINICAL TRIAL: NCT05078411
Title: Efficacy of Periodontal Risk Communication on Awareness and Propensity to Undergo the Suggested Treatments in Patients With and Without History of Tooth Loss Due to Periodontitis
Brief Title: Efficacy of Periodontal Risk Communication in Patients With and Without History of Tooth Loss
Acronym: PERIORISK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Leonardo Trombelli, Full Professor and Chair of Periodontology, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PERIORISK
Record Dates: First submitted 2021-09-17; First posted 2021-10-14 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis; Periodontal Diseases; Communication
Keywords: periodontitis; periodontal diseases; prognosis; risk assessment; risk factor; communication; consciousness; propensity
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Communication | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study is designed as a multicenter, single-blind, parallel-arm, randomized trial.
Who Masked: Outcomes Assessor
Masking Description: The examiner responsible for administrating psychological questionnaires will be kept blinded as to patient allocation to treatment (the examiner will leave the operating room when treatment allocation is disclosed and when the operator delivers the assigned treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without a history of tooth loss due to periodontitis (NTLP) (Other)
  Interventions: Behavioral: Test treatment; Behavioral: Control treatment
- Patients with a history of tooth loss due to periodontitis (TLP) (Other)
  Interventions: Behavioral: Test treatment; Behavioral: Control treatment

INTERVENTIONS:
Behavioral: Test treatment — Test treatment will consist of a single session structured as follows: (i) information on periodontal diagnosis (as formulated according to the classification system of the 2017 World Workshop for the Classification of Periodontal Diseases and Conditions); (ii) information on periodontal risk level (as calculated with the PerioRisk tool proposed by Trombelli et al. 2009) and profile (i.e., the magnitude of the contribution of each PerioRisk parameter to generate the patient risk level); (iii) information on treatment plan and oral hygiene instructions, with emphasis to treatment goals based on the PerioRisk output.
  The operators will be trained to administer test treatment in approximately 8 minutes, but the duration of the session will be extended for additional questions and answers upon patient request.
  Other Names: Periodontal risk assessment
Behavioral: Control treatment — Control treatment will consist in a single session structured as follows: (i) information on periodontal diagnosis (as formulated according to the classification system of the 2017 World Workshop for the Classification of Periodontal Diseases and Conditions); (ii) information on treatment plan and oral hygiene instructions, and treatment goals. Although the general concept of risk of periodontitis incidence/progression will be explained, no mention will be made to the patient risk level as calculated with PerioRisk or any other tool.
  The operators will be trained to administer control treatment in approximately 8 minutes, but the duration of the session will be extended for additional questions and answers upon patient request.
  Other Names: Treatment as usual

SUMMARY:
SCIENTIFIC BACKGROUND The periodontal risk assessment method proposed by the University of Ferrara (namely, the PerioRisk; Trombelli et al. 2009) has been retrospectively validated and has been shown as a promising tool for tailoring supportive periodontal care. No information on its efficacy on psychological outcomes, however, is currently available.

AIMS The primary aim of the study is to evaluate the efficacy of communicating periodontal risk level (as assessed with the PerioRisk tool) on psychological outcomes (i.e, patient consciousness and propensity to adhere to treatment instructions) in subjects who have been programmed for first periodontal consultation. The secondary aims of the study are (i) to comparatively evaluate the level of consciousness and propensity to adhere to treatment instructions in patients without a history of tooth loss due to periodontitis (as evaluated after communication of their periodontal risk level) and patients with a history of tooth loss due to periodontitis (as evaluated before their periodontal consultation); and (ii) to comparatively evaluate oral hygiene levels in patients who have received information on their diagnosis, treatment plan, oral hygiene instructions and treatment goals with or without the support of PerioRisk.

MATERIALS & METHODS Eighty patients (40 without a history of tooth loss due to periodontitis, NTLP; 40 with a history of tooth loss due to periodontitis, TLP) will be recruited at 2 centers and randomly assigned to receive test or control treatment. Therefore, each of the two treatment groups (test and control) will incorporate two subgroups (NTLP and TLP) of 20 patients each.

For each participant, the experimental phase of the study will consist of three observation intervals: T0 (verification of the eligibility criteria, patient allocation to treatment; T1 (performed within 3 months from T0 for assessment of clinical parameters, treatment administration, and administration of questionnaires before and after treatment; T2 (performed at 8-12 weeks after T1 for the assessment of clinical parameters).

At T1, following routine periodontal clinical assessment and questionnaire completion, patients will receive test or control treatment according to the randomization list. Test treatment will consist of a single session structured as follows: (i) information on periodontal diagnosis; (ii) information on periodontal risk level (as calculated with the PerioRisk tool) and profile (i.e., the magnitude of the contribution of each PerioRisk parameter to generate the patient risk level); (iii) information on treatment plan and oral hygiene instructions, with emphasis to treatment goals based on the PerioRisk output. Control treatment will consist in a single session structured as follows: (i) information on periodontal diagnosis; (ii) information on treatment plan and oral hygiene instructions, and treatment goals. Although the general concept of risk of periodontitis incidence/progression will be explained, no mention will be made to the patient risk level (as calculated with PerioRisk or any other tool) when administering control treatment. Two operators will be trained to administer test and control treatments in approximately 8', but time for treatment administration will be extended for additional questions and answers whenever needed by the patient. Total time for treatment administration will be recorded.

Patients will be administered the following battery of psychological questionnaires: (i) Positive Affect Negative Affect Scale (PANAS) (Watson et al. 1988); (ii) Protection Motivation Theory (PMT) questionnaire (Conner & Norman 2005); (iii) Hospital Anxiety and Depression Scale (HADS-A/D) (Zigmond & Snaith 1983). While HADS-A/D will be used to screen out patients with clinical anxiety/ depression before treatment administration, PANAS and PMT will be completed either immediately before and immediately after treatment administration.

DETAILED DESCRIPTION:
SCIENTIFIC BACKGROUND The standardized application of the same protocols (for intensity, modality, and monitoring) for primary and secondary prevention of periodontitis as well as for the active treatment phase itself will rarely meet the individual's needs, resulting in under-provision of care to some and over-provision to others, with unwanted side effects and suboptimal allocation of resources. To deliver personalized and precision periodontal care, risk assessment should be incorporated in the periodontal evaluation as a third dimension, to comprehensively assess and interpret factors that may have an impact on future disease onset or progression and upon a patient's anticipated response to periodontal treatment. Previous studies showed that patients receiving information on individual periodontal risk level had significantly higher consciousness of disease seriousness and significantly higher intention to adhere to treatment instructions after consultation. These findings support the use of this system in clinical practice and obtain greater patient adherence to the suggested preventive and treatment protocols. Although the periodontal risk assessment method proposed by the University of Ferrara (namely, the PerioRisk) has been retrospectively validated and has been shown as a promising tool for tailoring supportive periodontal care, no information on its efficacy on psychological outcomes is currently available.

AIM Primary aim: to evaluate the efficacy of communicating periodontal risk level (as assessed with the PerioRisk tool) on psychological outcomes (i.e, patient consciousness and propensity to adhere to treatment instructions) in subjects who have been programmed for first periodontal consultation.

Expected result (primary aim): when communicating information on periodontal diagnosis, periodontal treatment plan, oral hygiene instructions and periodontal treatment goals to the patient undergoing first periodontal consultation, the adjunctive use of the PerioRisk tool will result in significantly increased levels of patient consciousness and propensity to adhere to treatment instructions.

Secondary aim #1: to comparatively evaluate the level of consciousness and propensity to adhere to treatment instructions in (i) patients without a history of tooth loss due to periodontitis (as evaluated after communication of their periodontal risk level) and (ii) patients with a history of tooth loss due to periodontitis (as evaluated before their periodontal consultation).

Expected result (secondary aim #1): in subjects without a history of tooth loss due to periodontitis, the adjunctive use of the PerioRisk tool during first periodontal consultation will improve patient consciousness and propensity to adhere to treatment instructions up to levels that are reached with periodontitis-associated tooth loss.

Secondary aim 2: to comparatively evaluate oral hygiene levels in patients who have received information on their diagnosis, treatment plan, oral hygiene instructions and treatment goals with or without the support of PerioRisk during their consultation.

Expected result (secondary aim #2): at a distance of 8-12 weeks from consultation, greater improvements in full-mouth Plaque Index will be observed in patients who have received information on their diagnosis, treatment plan, oral hygiene instructions and treatment goals with the support of the PerioRisk tool.

EXPERIMENTAL DESIGN The study is designed as a multicenter, single-blind, parallel-arm, randomized trial.

MATERIALS & METHODS Participating clinical centers Participants will be recruited at 2 centers: (i) Section of Dentistry, University of Ferrara; and (ii) Operative Unit of Dentistry, Azienda Unità Sanitaria Locale of Ferrara, Italy.

Study population Specific inclusion and exclusion criteria will be used to recruit adult patients programmed for their first periodontal consultation. Patient selection will ensure a balanced distribution (1:1 ratio) of patients with and without a history of tooth loss due to periodontitis (Tooth Loss due to Periodontitis, TLP group; and No Tooth Loss due to Periodontitis, NTLP group).

Sample size Based on data from the study by Asimakopoulou et al. (2015), a per-protocol study of 62 patients will be sufficient to detect a significant inter-group difference in the primary outcome measure (i.e., patient propensity to adhere to treatment instructions) with a two-sided test at a p-level of 0.05 and a statistical power of 80%. An intention-to-treat population of 80 patients (40 allocated to test treatment, 40 allocated to control treatment) will be used for the study.

Observation intervals

For each participant, the experimental phase of the study will consist of three observation intervals:

T0 (screening visit): verification of the eligibility criteria, patient allocation to treatment; T1 (within 3 months from T0): assessment of clinical parameters; treatment administration; administration of questionnaires before and after treatment; T2 (8-12 weeks after T1): assessment of clinical parameters.

Experimental treatments and patient allocation to treatment Following routine periodontal clinical assessment and questionnaire completion (see study parameters for details), patients will receive test treatment (RISK) or control treatment (TaU) according to the randomization list (as created using a random digit generator). Before the study, two operators (A.S. and M.E.G.) will be trained to administer RISK or TaU in approximately 8 minutes. The patient will be left free to interrupt the session for questions, if needed. Only the operator and the patient will be present in the operating room during treatment administration. Whenever needed by the patient, time for treatment administration will be extended for additional questions and answers. Total time for treatment administration will be recorded.

Statistical methods Non-parametric two-sided statistical tests will be used for intra-group comparisons (i.e., pre- vs post-treatment administration; Wilcoxon paired samples test) and inter-group comparisons (i.e., RISK vs TaU and TLP vs NTLP; Mann-Whitney U-test) for scores obtained from the psychological questionnaires. Cronbach's alpha will be calculated for the PMT scale overall to assess internal consistency.

ELIGIBILITY:
Inclusion Criteria:

* possessing a recent (i.e., performed within 24 months) bidimensional radiograph (orthopantomography or periapical status) or programmed to perform the radiographic exam;
* speaking Italian fluently.

Exclusion Criteria:

* history of a previous periodontal diagnosis;
* conditions (es. psychiatric diseases, alcohol abuse) or drug exposures (e.g., antidepressants) that may influence the results of psychological questionnaires;
* lack of a recent (i.e., performed within 24 months) bidimensional radiograph and not able/willing to provide the exam (e..g., due to pregnancy);
* not presenting at two programmed study visits consecutively;
* pre-treatment HADS score indicative of clinical depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Propensity to adhere to treatment instructions over the next 8-12 weeks | up to 3 months following the screening visit (i.e., at T1, both before and after treatment administration)
  The outcome consists of the mean post-treatment change in the patient-related score related to the item "Intention" of the Protection Motivation Theory (PMT) questionnaire (Conner & Norman 2005). The score can range on a scale from 1 to 10, with higher scores indicating a better outcome (i.e., greater propensity to adhere to treatment instructions).

SECONDARY OUTCOMES:
Mean change in the score related to "Positive emotions" | up to 3 months following the screening visit (i.e., at T1, both before and after treatment administration)
  The outcome consists of the mean post-treatment change in the patient-related score related to the item "Positive emotions" of the Positive Affect Negative Affect Scale (PANAS) (Watson et al. 1988). The score can range on a scale from 10 to 50, with higher scores representing higher levels of positive affect.
Mean change in the score related to "Negative emotions" | up to 3 months following the screening visit (i.e., at T1, both before and after treatment administration)
  The outcome consists of the mean post-treatment change in the patient-related score related to the item "Negative emotions" of the Positive Affect Negative Affect Scale (PANAS) (Watson et al. 1988). The score can range on a scale from 10 to 50, with lower scores representing lower levels of negative affect.
Mean change in the score related to "Seriousness" | up to 3 months following the screening visit (i.e., at T1, both before and after treatment administration)
  The outcome consists of the mean post-treatment change in the patient-related score related to the item "Seriousness" of the Protection Motivation Theory (PMT) questionnaire (Conner & Norman 2005). The scores can range on a scale from 1 to 10, with higher scores indicating a better outcome.
Mean change in the score related to "Susceptibility" | up to 3 months following the screening visit (i.e., at T1, both before and after treatment administration)
  The outcome consists if the mean post-treatment change in the patient-related score related to the item "Susceptibility" of the Protection Motivation Theory (PMT) questionnaire (Conner & Norman 2005). The scores can range on a scale from 1 to 10, with higher scores indicating a better outcome.
Mean change in the score related to "Treatment effectiveness" | up to 3 months following the screening visit (i.e., at T1, both before and after treatment administration)
  The outcome consists of the mean post-treatment change in the patient-related score related to the item "Treatment effectiveness" of the Protection Motivation Theory (PMT) questionnaire (Conner & Norman 2005). The scores can range on a scale from 1 to 10, with higher scores indicating a better outcome.
Mean change in the score related to "Self-efficacy" | up to 3 months following the screening visit (i.e., at T1, both before and after treatment administration)
  The outcome consists if the mean post-treatment change in the patient-related score related to the item "Self-efficacy" of the Protection Motivation Theory (PMT) questionnaire (Conner & Norman 2005). The scores can range on a scale from 1 to 10, with higher scores indicating a better outcome.
Mean change in the score related to "Treatment barriers" | up to 3 months following the screening visit (i.e., at T1, both before and after treatment administration)
  The outcome consists of the mean post-treatment change in the patient-related score related to the item "Treatment barriers" of the Protection Motivation Theory (PMT) questionnaire (Conner & Norman 2005). The scores can range on a scale from 1 to 10, with lower scores indicating a better outcome.
Mean change in the score related to "Fear" | up to 3 months following the screening visit (i.e., at T1, both before and after treatment administration)
  The outcome consists of the mean post-treatment change in the patient-related score related to the item "Fear" of the Protection Motivation Theory (PMT) questionnaire (Conner & Norman 2005). The scores can range on a scale from 1 to 10, with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Operative Unit of Dentistry, Azienda Unità Sanitaria Locale (AUSL), Ferrara
  - Section of Dentistry, University of Ferrara, Ferrara

REFERENCES:
- [Derived] Farina R, Simonelli A, Guarnelli ME, Secchiati G, Montemezzo G, Scapoli C, Trombelli L. Efficacy of communicating periodontal risk on psychological outcomes and supragingival plaque control in patients undergoing first periodontal consultation: A parallel-arm, randomized trial. J Clin Periodontol. 2024 Oct;51(10):1289-1301. doi: 10.1111/jcpe.14032. Epub 2024 Jul 2. PMID 38956317